CLINICAL TRIAL: NCT00176085
Title: Pharmacokinetics of 11-Nor-9-carboxy-D9-tetrahydrocannabinol (THCCOOH) and Its Acyl-glucuronide (THCCOOH-GLu) After Intravenous Administration of THCCOOH in Healthy Human Subjects
Brief Title: Pharmacokinetics of THCCOOH and Its Acyl-glucuronide After Intravenous Administration of THCCOOH
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Other Study IDs: K107
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: THCCOOH; Pharmacokinetics; Metabolism; Cannabis
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- healthy: healthy volunteers

SUMMARY:
A study on the fate and elimination of 11-Nor-Delta9-carboxy-9-tetrahydrocannabinol was up to now not conducted, except of one single experiment in which (lacking) psychopharmacological activity was tested after intravenous infusion of 20 mg in a human individual. In this study, however, the authors did not trace the above questions due to analytical and methodological deficits.

Aim of the study is to determine the pharmacokinetics of THCCOOH and THCCOOH-Glu after intravenous ad-ministration of 5 mg THCCOOH in healthy individuals

DETAILED DESCRIPTION:
To determine the pharmacokinetics of THCCOOH after intravenous administration of THCCOOH (5 mg) and its formed glucuronide in healthy individuals in order to improve the possibilities for the assessment of unfitness to drive. For these purposes the following criteria will be studied:

THCCOOH

* Primary: Area under the plasma concentration time curve (AUCtotal) Maximal plasma concentrations (Cmax) Time of Cmax (tmax) Terminal elimination half-life (t1/2)
* Secondary: Systemic and renal clearance (Cls, CLr) Volume of distribution of (Vc) Formed THCCOOH-glu
* Primary: Area under the plasma concentration time curve (AUCtotal) Maximal plasma concentrations (Cmax) Time of Cmax (tmax) Terminal elimination half-life (t1/2)
* Secondary: Systemic and renal clearance (Cls, CLr) Volume of distribution (Vc)

ELIGIBILITY:
Inclusion Criteria:

* Good state of health (physically and mentally)

Exclusion Criteria:

* Any regular drug treatment within the last two months
* Any intake of a substance known to induce or inhibit drug metabolising enzymes or transport systems within a period of less than 10 times the respective elimination half-life
* Any acute or chronic illness or clinically relevant findings in the pre-study examination
* Allergies (except for mild forms of hay fever) or history of hypersensitivity reactions
* Smoking (regular or irregular)
* Excessive alcohol drinking (more than approximately 30 g alcohol per day)
* Positive drug screening especially THC or known or admitted drug abuse

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 2004-10; Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Mikus, MD BSc, Principal Investigator — Department of Internal Medicine VI
Locations (1):
- Clinical Research Center, Department of Internal Medicine VI, Heidelberg, Germany